CLINICAL TRIAL: NCT02249611
Title: Application of Mobile Physical Activity Promotion Tool in Subjects With Overweight/Metabolic Abnormality---randomised Control Trial of Efficacy
Brief Title: Application of MT in Subjects With Overweight/Metabolic Abnormality---RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Yi-Ching Yang, MD, professor, National Cheng-Kung University Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: NSC 102-2314-B-006 -004 -MY2
Record Dates: First submitted 2014-09-23; First posted 2014-09-25 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Overweight; Metabolic Abnormality
Keywords: Physical activity; mobile activity sensor and feedback system; self-management of health
MeSH Terms: conditions — Overweight; Motor Activity | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MT and life counseling (Experimental): To improve physical activity, body composition, physiological parameters and quality of life by using MT (mobile physical activity promotion tool) and lifestyle counseling in diet control, increased physical activity, less smoking and drinking, deal with pressure, and regular health examination will be conducted for 3 months in intervention periods.
  Interventions: Device: Mobile physical activity promotion tool
- Standard care (Active Comparator): Lifestyle counseling in diet control, increased physical activity, less smoking and drinking, deal with pressure, and regular health examination based on the booklet of metabolic syndrome prevention which is edited by Health Promotion Administration, Ministry of Health and Welfare in Taiwan only once in this period (3 months).
  Interventions: Other: Standard care

INTERVENTIONS:
Device: Mobile physical activity promotion tool — 1. Mobile activity sensor
  2. Smartphone with APP
  3. Interactional webpage of internet
  4. Evidence based health information
  5. Individualized reminding messages according to the data from activity recording system
  6. Personal counseling from professional personnel
  Arms: MT and life counseling
Other: Standard care — Counseling on lifestyles with health education material
  Other Names: Counseling on lifestyles
  Arms: Standard care

SUMMARY:
The subjects will be recruited from July 1, 2014 until the participants enough. Interviewing for research purpose explication and informed consent will be collected before the study is executed. In the first 3 months, subjects of group A will use the mobile physical activity promotion tool (MT), receive professional personal counseling, and individualized reminding message (intervention) once a week. In the last 3 months, they will receive standard care (control) which is in support of behavioral and educational recommendations in diet control, increased physical activity, less smoking and drinking, deal with pressure, and regular health examination (based on the booklet of metabolic syndrome prevention which is edited by Health Promotion Administration, Ministry of Health and Welfare, Taiwan). Subjects of group B will begin with an initial 3 months control period of standard care only, and the intervention program will be conducted for last 3 months.

DETAILED DESCRIPTION:
RCT with a crossover design will present in this study and take place during a 6-month period. Participants will be randomly allocated to two groups applying a randomized block technique and matching with different age and sex. The subjects will be recruited from July 1, 2014 until the participants enough. Interviewing for research purpose explication and informed consent will be collected before the study is executed. Physical activity amount (including mild, moderate and vigorous physical activity), cardio-respiratory fitness (including three minutes of stair-climbing and a minute sit-up), physiological indicators (blood pressure, weight, waist circumference, and body composition), metabolic and biochemical indicators (including glucose level, lipid profile etc.), and the questionnaire of psychological health and quality of life will be recorded at the first visit. And then subjects will be followed after 12 weeks and 24 weeks. Additionally, diet record compliance will be recorded for 12 weeks.

In the first 3 months, subjects of group A will use the mobile physical activity promotion tool (MT), receive professional personal counseling, and individualized reminding message (intervention) once a week. In the last 3 months, they will receive standard care (control) which is in support of behavioral and educational recommendations in diet control, increased physical activity, less smoking and drinking, deal with pressure, and regular health examination (based on the booklet of metabolic syndrome prevention which is edited by Health Promotion Administration, Ministry of Health and Welfare, Taiwan). Subjects of group B will begin with an initial 3 months control period of standard care only, and the intervention program will be conducted for last 3 months.

ELIGIBILITY:
Inclusion criteria:

* Body Mass Index (BMI) ≥ 24kgw/m2,
* Waist circumference, male≥ 90cm, female≥ 80cm,
* Systolic blood pressure ≥ 130 mmHg or diastolic blood pressure ≥ 85mmHg,
* Fast plasma glucose ≥ 100mg/dL,
* High-density lipoprotein cholesterol (HDL-C): male<40 mg/dL, female<50 mg/dL,
* Triglyceride ≥ 150 mg/dL.

Exclusion criteria:

* can't use computer, internet, and smartphone,
* is pregnant, within 6 months after delivery and on breastfeeding,
* is exercise-intolerance.
* use the relevant drugs for weight reduction, cardiovascular diseases, hypertension, diabetes and dyslipidemia.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2014-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Increase physical activity | 6 months
  Measurement by mobile activity sensor system and the questionnaire of International Physical Activity Questionnaires (IPAQ) short form, and evaluate by counts/minute

SECONDARY OUTCOMES:
Increase physical fitness | 6 months
  Measurement by examination of physical fitness.

OTHER OUTCOMES:
executive performance of participants | 6 months
  physiological indicators and other metabolic and biochemical indicators, the questionnaire of psychological health, and WHO health related quality of life to evaluate executive performance of participants
diet record compliance | 3 months
  Measurement by records of web survey

CONTACTS AND LOCATIONS:
Overall Officials: Yi Ching Yang, MD, Principal Investigator — Department of Family Medicine, College of Medicine, National Cheng Kung University
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

REFERENCES:
- [Derived] Yang YP, Wang CJ, Wang JJ, Lin CW, Yang YC, Wang JS, Yang YK, Yang YC. The Effects of an Activity Promotion System on active living in overweight subjects with metabolic abnormalities. Obes Res Clin Pract. 2017 Nov-Dec;11(6):718-727. doi: 10.1016/j.orcp.2017.06.002. Epub 2017 Jul 17. PMID 28729003